CLINICAL TRIAL: NCT01210703
Title: Evaluation of Effect of Continuous Positive Air Pressure (CPAP) on Upper Airway Dimensions, by Acoustic Pharyngometry (AP), in Severe Obstructive Sleep Apnea Syndrome (OSAS) and Primary Snore Patients
Brief Title: Acoustic Pharyngometry in Obstructive Sleep Apnea Syndrome Patients, With Indication of Continuous Positive Air Pressure
Acronym: APOSAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Luiz Ubirajara Sennes, University of Sao Paulo General Hospital
Other Study IDs: AcPh.1
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Acoustic Pharyngometry; CPAP; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Acoustic Pharyngometry (AP) is a method of measurement of Transversal Sectional Areas (TSA) and Volumes of oral cavity and pharynx, based on acoustic waves. The aim of this study is to describe changes on oropharynx dimensions caused by CPAP (Continuous Positive Air Pressure) in patients with severe Obstructive Sleep Apnea Syndrome when compared with patients with Primary Snore, using AP. The exam will be made during the use of CPAP, at various pressures. The investigators also intend to determine if pressure determined by Polysomnography in OSAS patients cause some type of different change in AP graphic.

DETAILED DESCRIPTION:
The investigators are performing AP exams in severe apneics (cases) and primary snorers (control group),first basal, and then at the same time of using CPAP with a nasal mask, at progressive pressures (from 4 to 10 cmH20 in snorers, and until 2 pressures above the polysomnography determined pressure in apneics). The wave tube of pharyngometer is connected to the patient´s mouth by a mouthpiece, and to the computer. It makes a graphic of area x distance for each measurement. Then the investigators compare the changes in area, distance and volume of oral cavity and pharynx, determined by CPAP pressures, in both groups, and compare the measurements inside each group and between the two groups. Finally, the investigators analyse the CPAP pressure that most modifies the AP graphic, observing if it has some relationship with the polysomnography determined CPAP pressure.

The investigators intend this way to show the kind of modifies determined by CPAP in oral cavity and oropharynx and, secondarily, observe some relationship of AP and polysomnography in determine the CPAP ideal pressure for severe apneic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old
* Female and male

Exclusion Criteria:

* Cardiopathies
* Chronic nasal obstruction
* Using neurologic or psychiatric drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Severe Sleep Obstructive Apnea Syndrome and Primary Snorers, who have already made a polysomnography (in apneics, polysomnography for CPAP titulation, too).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Inês G de Sousa Silva, Md, Principal Investigator — University of São Paulo General Hospital; Luiz U Sennes, Phd, Study Director — University of Sao Paulo General Hospital; Michel B Cahali, Phd, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Otolaringology Ambulatory of University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil